CLINICAL TRIAL: NCT00163111
Title: A Randomized, Open Label, Comparative Multicenter Study Of Voriconazole Versus Conventional Amphotericin B Followed By Fluconazole In The Treatment Of Candidaemia In Non Neutropenic Subjects.
Brief Title: A Clinical Study Intended To Compare Treatment With Voriconazole To Treatment With Amphotericin Followed By Fluconazole In Patients With Candidemia, A Serious Fungus Infection Of The Blood.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 608; A1500608
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis

INTERVENTIONS:
Drug: VFENDÂ® I.V., Oral
Drug: Conventional amphotericin B
Drug: Diflucan IV, oral

SUMMARY:
This is a study to investigate the safety and efficacy of voriconazole for the treatment of candidemia in critically ill non-neutropenic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with candidemia

Exclusion Criteria:

* Neutropenia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 1998-09; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Sustained clinical response for 12 weeks from end of treatment

SECONDARY OUTCOMES:
Time to negative blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer